CLINICAL TRIAL: NCT01150682
Title: Role of Sex Hormone and Insulin/IGF Axes in Endometrial Cancer Recurrence
Brief Title: Role of Biomarkers in Endometrial Cancer Recurrence in Samples From Patients With Stage II, Stage III, or Stage IV Endometrial Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Philip J. DiSaia, Gynecologic Oncology Group
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000680598; GOG-8015
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2010-08

CONDITIONS: Endometrial Cancer
Keywords: endometrial adenocarcinoma; stage II endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; endometrial adenosquamous cell carcinoma; endometrial clear cell carcinoma; endometrial papillary serous carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Reverse Transcriptase Polymerase Chain Reaction; Enzyme-Linked Immunosorbent Assay; Immunohistochemistry

INTERVENTIONS:
Genetic: RNA analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: enzyme-linked immunosorbent assay
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research study is studying the role of biomarkers in endometrial cancer recurrence in samples from patients with stage II, stage III, or stage IV endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the association of endometrioid adenocarcinoma (EA) recurrence with pre-operative serum levels of insulin, total and free insulin-like growth factor-I (IGF-I), IGF-II, insulin-like growth factor-binding protein-1 (IGFBP-1) and IGFB-3, estradiol, estrone, progesterone, and sex hormone-binding globulin (SHBG) in samples from patients with stage II-IV endometrial cancer evaluated on GOG-0210.
* To study the associations of EA recurrence with pre-treatment tumor expression of IGF-I, IGF-II, and IGFBP-1 and -3 mRNA in samples from these patients.
* To study the associations of EA recurrence with pre-treatment tumor expression of insulin receptor, IGF-I receptor, estrogen receptor, and progesterone receptor in samples from these patients.
* To measure the correlations of serum (protein) and tissue (mRNA) levels of IGF-I, IGF-II, and IGFBP-1 and -3 from samples of patients with EA and participants without cancer.

OUTLINE: Banked serum and tumor tissues samples are analyzed for levels of insulin, total and free insulin-like growth factor (IGF-I), IGF-II, IGFBP-1 and IGFBP-3, estradiol, estrone, progesterone and sex hormone-binding globulin (SHBG); expression of IGF-I, IGF-II, IGFBP-1 and IGFBP -3 mRNA; and expression of the insulin receptor, IGF-I receptor, estrogen receptor, and progesterone receptor by RT-PCR, IHC, and ELISA. Banked non-cancerous endometrial tissue and fasting serum samples from controls are also analyzed for IGF-I, IGF-II, IGFBP-1, and IGFBP-3 and compared with the results of endometrial adenocarcinoma (EA) samples.

Clinical information associated with each EA samples (i.e., age, BMI, performance status, race, ethnicity, tumor stage, size, histology and grade, surgical compliance and type of post surgical adjuvant therapy, overall survival, recurrence-free survival, site of first recurrence, and biomarker values and expression) is also collected.

PROJECTED ACCRUAL: A total of 815 patient specimens and 50 control specimens will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed endometrioid endometrial cancer

  * Stage II-IV disease
* Patients who were eligible and evaluated on the GOG-0210, Molecular Staging in Endometrial Cancer clinical trial, meeting the following criteria:

  * Allowed their specimens and clinical data collected as part of their participation
  * Have sufficient high-quality frozen primary tumor, formalin-fixed and paraffin-embedded (FFPE) primary tumor, and/or pre-operative serum for testing available
* Patients who underwent surgical staging as specified in the GOG-0210 protocol and described in the GOG Surgical Manual Protocol, including any of the following procedures:

  * Hysterectomy
  * Bilateral oophorectomy
  * Washings as well as pelvic lymphadenectomy and para-aortic lymphadenectomy
* Non-cancerous endometrial tissue and fasting serum from control samples meeting the following criteria (controls):

  * Underwent hysterectomy to treat uterine prolapse at the Albert Einstein Hospital and Montefiore Medical Center, in the Bronx, NY
  * No uterine fibroids or prior cancer

PATIENT CHARACTERISTICS:

* Postmenopausal patients and controls

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 865 (Estimated)
Dates: Start 2010-07; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Patient characteristics: age, BMI, performance status, race, ethnicity
Tumor characteristics
Surgical compliance and type of surgical adjuvant therapy
Overall survival
Recurrence-free survival
Site of first recurrence
Biomarker values and expression levels

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gunter, PhD, Principal Investigator — Albert Einstein College of Medicine